CLINICAL TRIAL: NCT03754699
Title: Impact of a Preoperative Education on the Quality of Postoperative Analgesia Management in Outpatient Surgery
Brief Title: Preoperative Education for Less Outpatient Pain After Surgery (PELOPS)
Acronym: PELOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL17_0860; 2018-A00010-55 (Other: ANSM)
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Outpatient Orthopedic Surgery
Keywords: Pain; Surgery; Preoperative Education; Outpatient
MeSH Terms: conditions — Pain | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with a therapeutic educational intervention (Experimental): Arm 1 : Interventional group: A therapeutic educational intervention is performed following pre-anesthesia assessment
  Interventions: Behavioral: Educational intervention
- Patients without therapeutic educational intervention (Active Comparator): Arm 2 : Control group: standard information on pain is performed following pre anesthesia assessment
  Interventions: Behavioral: Standard information

INTERVENTIONS:
Behavioral: Educational intervention — During the usual pre-anesthesia assessment (performed between D-30 and D0 of the intervention), the anesthesiologist will deliver to the intervention group patient oral and visual information on:
  * the numerical scale of pain ranging from 0 to 10 with examples of perceptions corresponding to each level of the scale (calibration)
  * nature of postoperative pain (inflammatory character, dynamic over time)
  * average pain level incurred by the intervention
  * the difference between anti-inflammatory and opioid analgesics
  * principles of systematic treatment and pain anticipation
  * principles of overdose and side effects prevention This information is standardized and delivered orally, accompanied by a visual support (patient diary), which will be given to the patient upon discharge from the hospital
  Arms: Patients with a therapeutic educational intervention
Behavioral: Standard information — Standard information on pain For patients in the control group the standardized information is based on the SG/DGM/DSS 1/41-2010 scheme of the AFSSAPS-CFETD repository.
  Arms: Patients without therapeutic educational intervention

SUMMARY:
In 2015, more than 50% of surgical procedures were performed in outpatient settings. Successful pain management after outpatient surgery is crucial, and requires a perfect cooperation between caregivers and patients, with clear information on the analgesics use at home. Different strategies to control postoperative pain were adopted by hospitals performing outpatient surgery. However, up to half of patients receive little or no information about the treatment of postoperative pain, and at least one third of them are not able to follow postoperative analgesia instructions. There is a clear unmet need in pain treatment during first 48-72 hours after discharge, with important number of emergency calls and readmissions. The most common causes of rescue calls after outpatient surgery are uncontrolled pain and questions about medications or post-operative care.

Structured education interventions using psychological techniques to enhance engagement and behavior were found to be beneficial for better acute pain management in outpatient settings after orthopedic surgery.

We hypothesize that an educational intervention based on the rational perception of postoperative pain and discomfort, and the proper use of analgesics would improve the quality of pain management at home and reduce analgesics-related side effects.

Principal objective of this study is to evaluate the impact of a preoperative educational intervention on effectiveness of postoperative pain self-management in outpatient settings compared to the current practice.

Secondary objectives are to evaluate the prevalence of analgesics use and the incidence of severe pain episodes, as well as side effects. The occurrence of neurological pain, quality of sleep, and patient's comfort will be evaluated at 30th day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years);
* Patients scheduled for outpatient orthopedic surgery
* ASA (American Society of Anesthesiology) I to III;
* Patients admitted for an outpatient intervention resulting in moderate to severe pain: eg: arthroscopy of the knee or shoulder, cruciate ligaments, shoulder block, medial patellofemoral ligament plasty (not exhaustive)

Exclusion Criteria:

* Pregnant or lactating women
* Patients with contraindications to paracetamol and/or second-level analgesic and/or NSAIDs (hepatocellular insufficiency, respiratory insufficiency, substituted or unsubstituted drug addicts, allergy to one of the drugs, history of bleeding or digestive perforation during previous NSAID treatment, history of gastroduodenal ulcer, renal failure with clearance <50mL / min, severe heart failure)
* Patients with preoperative chronic pain (outside operative site, known or detected by DN4)
* Patients admitted for an outpatient arthroplasty (excluded because they are subjected of a specific preoperative preparation)
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care, persons admitted to a health or social establishment for other purposes than research
* Patient with a poor understanding of French
* Patient refusing to participate to the study
* Patient not affiliated to a social security regimen
* Patient participating in other interventional research except a routine care research (former regulation) and/or research with no interference with the primary endpoint analysis as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Time-weighted sum of Pain Relief - Total Pain Relief (TOTPAR) during 5 postoperative days | Day 5
  TOTPAR is a global score based on relief of pain. A numerical scale has at its left end the words "no relief = 0" and at its right end "complete relief = 100%". The pain relief score is calculated using the area under the curve for a defined period of time. TOTPAR is also expressed as a percentage of the maximum TOTPAR that would be achieved by treatment that would provide complete relief during the observation period. In order to measure this area under the curve, at least 3 measurements per day will have to be reported in the patient diary.

SECONDARY OUTCOMES:
Time-weighted sum of Pain Relief - Total Pain Relief (TOTPAR) | At Day 10, Day 20 and Day 30 with the initial point at Day 5
  TOTPAR is a global score based on relief of pain. A numerical scale has at its left end the words "no relief = 0" and at its right end "complete relief = 100%". The pain relief score is calculated using the area under the curve for a defined period of time. TOTPAR is also expressed as a percentage of the maximum TOTPAR that would be achieved by treatment that would provide complete relief during the observation period. In order to measure this area under the curve, at least 3 measurements per day will have to be reported in the patient diary.
Type, number and doses of prescribed analgesics | At Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 10, Day 20 and Day 30.
  Patient will report drug intake on a patient diary
Incidence of severe pain (≥ 7 out of 10). | From day 0 to the end of stidy (Day 30)
  The patient diary will provide a continuous assessment at home of the pain intensity
Incidence of side effects (nausea / vomiting / gastralgia / dizziness / concentration disorder / somnolence / constipation, other). | From day 0 to the end of stidy (Day 30)
  Side effects will be collected on the patient diary
Prevalence of neuropathic pain assessed by using the DN4 scale. | At Day 30
  Patient will complete the DN4 questionnaires the day of the pre-anesthetic consultation and at Day 30 on the patient diary.
Sleep quality at day 0 and day 30 by the Pittsburgh Sleep Quality Index | At Day 0 and Day 30
  Patient will complete the PSQI questionnaires the day of the pre-anesthetic consultation and at Day 30 on the patient diary.
Comfort and experience of the patient evaluated by the International Pain Outcome questionnaire. | At Day 30
  Patient will complete the International Pain Outcome questionnaire at day 30, on the patient diary

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse - Anaesthesia Reanimation unit, Lyon, France

REFERENCES:
- [Derived] Dziadzko M, Bouteleux A, Minjard R, Harich J, Joubert F, Pradat P, Pantel S, Aubrun F. Preoperative Education for Less Outpatient Pain after Surgery (PELOPS trial) in orthopedic patients-study protocol for a randomized controlled trial. Trials. 2022 May 21;23(1):422. doi: 10.1186/s13063-022-06387-6. PMID 35598000